CLINICAL TRIAL: NCT05790083
Title: Assessment of the Short- and Long-Term Skin Efficacy and Tolerability of a Cosmetic Product Combination of Body Lotion and Intensive Care Over 3 Months in Subjects With Atopic Eczema
Brief Title: Skin Efficacy and Tolerability of a Cosmetic Product Combination Over 3 Months in Subjects With Atopic Eczema
Acronym: AtoCare-OS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bionorica SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AtoCare-OS
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Atopic Dermatitis; Eczema-Prone Skin
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Critical Care

STUDY DESIGN:
Masking Description: Trade name of products was masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body Lotion BNO 3732 + Intensive Care BNO 3731 (Experimental)
  Interventions: Other: Body Lotion and Intensive Care

INTERVENTIONS:
Other: Body Lotion and Intensive Care — Body Lotion, applied twice daily on whole body, for 3 months. Intensive Care, applied as needed on affected body areas.

SUMMARY:
The aim of this exploratory study is to investigate the short- and long-term efficacy and tolerability of a cosmetic product combination consisting of a body lotion and an intensive care product in subjects with atopic eczema over 3 months of use. Efficacy is assessed by instrumental measurements of skin condition (sub-panel), clinical examinations, and questionnaires.

DETAILED DESCRIPTION:
The objective of this exploratory study is to investigate the short- and long-term efficacy and tolerability of a cosmetic product combination consisting of a body lotion and an intensive care product in subjects with atopic eczema over 3 months of use.

For efficacy and tolerability evaluation, an objective dermatological assessment will be performed, in addition to assessing efficacy, the severity of atopic eczema will be assessed using the validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD). Further, the effect of the test product combination on symptom severity, disease control (recap of atopic eczema (RECAP)), quality of life and well-being will be evaluated by the subjects or the subjects' parents/ legal guardians. The subjects or the subjects' parents/ legal guardians will also document the frequency of flare-ups, required physician visits and the use of cortisone administration as well as their/ their child's well-being in a diary.

Additionally, the influence of the test product combination on the skin barrier will be assessed in a sub-panel with dry legs by measuring the transepidermal water loss by Aquaflux and by sampling of biological material for analysis of skin lipids and corneocyte maturity before and after 3 months of product use.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent of the subject to participate in the study, or, for underaged subjects of the parents/ legal guardians to let their child participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits or, for underaged subjects, willingness of the parents/ legal guardians to actively support their child's participation in the study and to come to the scheduled visits with their child
* Female and/or male
* Children from 2 to 17 years of age and adult subjects between 18 and 75 years of age
* Eczema-prone skin and atopic dermatitis, diagnosed by the dermatologist

Exclusion Criteria:

* Female subjects (only of childbearing age): Pregnancy or lactation
* Drug addicts, alcoholics (only adults)
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* Insulin-dependent diabetes mellitus
* One of the following illnesses with reduced physical capability/fitness: asthma (symptom-free allergic asthma is not an exclusion criterion), hypertension, cardiovascular diseases
* Documented allergies to cosmetic products and/or ingredients, skin care and/ or skin cleansing products as well as to ingredients of the test products
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, etc. at the test area that could influence the investigation
* Systemic therapy with immuno-suppressive drugs (e.g. corticosteroids, cyclosporine, dupilumab) and/or antihistamines (e.g. antiallergics) within the last 7 days prior to the start of the study
* Systemic therapy with anti-phlogistic agents or analgetics (e.g. diclophenac, ibuprofen), except for minor pain relief medicine like acetylsalicylic acid or paracetamol within the last 3 days prior to the start of the study
* Any topical medicinal products (e.g. topical corticosteroids, calcineurin inhibitors) at the test area within the last 5 days prior to the start of the study
* Any topical medication at the test area throughout the entire course of the study (except the medication normally used for treatment of atopic eczema)

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in objective dermatological evaluation of skin status (erythema, dryness, scaling, fissures, papules, pustules, edema, vesicles, weeping) by dermatologist (min = 0, max = 3; 3 = worst outcome) to Day 29, Day 57 and Day 85 | 85 days of treatment
Change from baseline in Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-ADTM, (min = 0, max = 3; 3 = worst outcome) to Day 29, Day 57 and Day 85 | 85 days of treatment
Change from baseline in Recap of atopic eczema (RECAP, min = 0, max = 4; 4 = worst outcome) to Day 29, Day 57 and Day 85 | 85 days of treatment
Change from baseline in Dermatology Life Quality Index (DLQI, 10 closed questions with varying scales) to Day 29, Day 57 and Day 85 | 85 days of treatment

SECONDARY OUTCOMES:
Change from baseline in the scoring of subjective dermatological evaluation via questionnaire (adults) (no scales) to Day 29, Day 57 and Day 85 | 85 days of treatment
Evaluation of product traits via questionnaire (7 questions with different answers, no scales) on day 1 and after 29, 57, 85 days | 85 days of treatment
Sub-group: mean change from baseline in transepidermal water loss (g/m2h), Lipid contents (ng/133mm²) and Morphological analysis (length of lipid lamellae, nm/1.000nm²) to Day 85 | 85 days of treatment
Safety of BNO 3732 and BNO 3731 measured by reported Adverse Events to Day 85 | 85 days of treatment
Subject diary (frequency of flare-ups, required physician visits, required drug administration/use of cortisone, well-being) | 85 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Unbereit, Dr., Principal Investigator — proDERM GmbH
Locations (1):
- SGS proderm GmbH, Schenefeld, Germany